CLINICAL TRIAL: NCT07335029
Title: Investigation of Hemodynamics and Radiomics Based on High Resolution Magnetic Resonance Imaging for Predicting the Outcomes of Intracranial Dissecting Aneurysm
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Principal Investigator, Li wenqiang, Doctor, Beijing Neurosurgical Institute
Other Study IDs: KY2024-315-02
Record Dates: First submitted 2026-01-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cerebrovascular Disease; Intracranial Aneurysm; Intracranial Arterial Dissection
MeSH Terms: conditions — Cerebrovascular Disorders; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group (Non-progression Group): Imaging progression of intracranial dissecting aneurysms during follow-up
- Experimental Group (Progression Group): Imaging progression of intracranial dissecting aneurysms during follow-up

SUMMARY:
This study aims to conduct a comprehensive analysis by integrating clinical factors, aneurysm morphological characteristics, and factors reflecting pathophysiological processes (such as hemodynamic and radiomics features), in order to explore the hemodynamic mechanisms associated with the progression of intracranial dissecting aneurysms. Furthermore, artificial intelligence algorithms will be employed to develop and validate an intelligent risk prediction model for the progression and outcomes of intracranial dissecting aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Intracranial dissecting aneurysm clearly diagnosed by DSA and high-resolution MRI imaging (according to the imaging diagnostic criteria proposed in the Chinese Expert Consensus on Imaging Diagnosis of Intracranial Arterial Dissection)
2. patients managed with conservative treatment and follow-up
3. patients who agree and sign a written informed consent form

Exclusion Criteria:

1. Arteritis, fibromuscular dysplasia, iatrogenic or traumatic pseudoaneurysms
2. Contraindications to MRI examination (such as claustrophobia or metallic implants), or contraindications to cerebral angiography (such as iodine contrast allergy)
3. Dissecting aneurysms extending from the extracranial segment to the intracranial segment, or cases with concomitant intracranial atherosclerotic plaques in the affected vessels
4. Patients who refuse MRI examination
5. Patients with severe comorbid diseases and an expected survival time of less than 2 years due to these conditions
6. Patients without follow-up HR-MRI imaging for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of patients with intracranial artery dissection (IAD) who received care at the study institution between 2015 and 2025. Eligible participants are adults aged 18-80 years with IAD confirmed by both digital subtraction angiography (DSA) and high-resolution MRI (HR-MRI) according to the imaging diagnostic criteria proposed in the Chinese expert consensus on intracranial artery dissection. Participants are managed with conservative treatment and undergo follow-up, and they provide written informed consent. Key exclusions include arteritis, fibromuscular dysplasia, iatrogenic or traumatic pseudoaneurysm; contraindications to MRI or cerebral angiography (e.g., implanted metallic foreign bodies, claustrophobia, or iodinated contrast allergy); extracranial dissection extending intracranially or concomitant intracranial atherosclerotic plaque in the affected vessel; refusal of MRI; severe comorbidities with an expected survival of less than 2 years; or absence of
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression of intracranial dissecting aneurysms | From enrollment to 12 months of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, the decision was made not to share the data.

REFERENCES:
- [Result] Li W, Liu J, Zhang Y, Wang K, Tian Z, Zhang Q, Jiang C, Yang X, Wang Y. Flow Diversion and Outcomes of Vertebral Fusiform Aneurysms After Stent-Only Treatment: A Hemodynamic Study. World Neurosurg. 2017 Nov;107:202-210. doi: 10.1016/j.wneu.2017.07.157. Epub 2017 Aug 4. PMID 28826706
- [Result] Zhang Y, Tian Z, Zhu W, Liu J, Wang Y, Wang K, Zhang Y, Yang X, Li W. Endovascular treatment of bilateral intracranial vertebral artery aneurysms: an algorithm based on a 10-year neurointerventional experience. Stroke Vasc Neurol. 2020 Sep;5(3):291-301. doi: 10.1136/svn-2020-000376. Epub 2020 Aug 13. PMID 32792460